CLINICAL TRIAL: NCT01396161
Title: A Phase 1 Placebo-controlled Study To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Ascending Oral Doses Of Pf-05175157 In Healthy Volunteers And In Patients With Type 2 Diabetes Mellitus (t2dm)
Brief Title: A Study of PF-05175157 in Healthy Volunteers and Type 2 Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Basic Science
Other Study IDs: B1731007
Record Dates: First submitted 2011-06-20; First posted 2011-07-18 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Phase 1; Multiple Doses; Safety; Pharmacokinetics; Pharmacodynamics; Healthy Volunteers; Type 2 Diabetic Patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 30 mg PF-05175157 or Placebo QD (Experimental)
  Interventions: Drug: PF-05175157 or Placebo
- 100 mg PF-05175157 or Placebo QD (Experimental): Planned dose might be modified based on emerging safety and PK data.
  Interventions: Drug: PF-05175157 or Placebo
- 200 mg PF-05175157 or Placebo QD (Experimental): Planned dose might be modified based on emerging safety and PK data.
  Interventions: Drug: PF-05175157 or Placebo
- 100 mg PF-05175157 or Placebo BID (Experimental): Planned dose might be modified based on emerging safety and PK data.
  Interventions: Drug: PF-05175157 or Placebo
- xxx mg PF-05175157 (Experimental): Dose will be determined based on results obtained from Arms 1 to 4.
  Interventions: Drug: PF-05175157 or Placebo

INTERVENTIONS:
Drug: PF-05175157 or Placebo — One oral dose of PF-05175157 or placebo is administered as a powder-in-capsule once daily for 14 days immediately before breakfast, in healthy volunteers.
  Arms: 30 mg PF-05175157 or Placebo QD
Drug: PF-05175157 or Placebo — One oral dose of PF-05175157 or placebo is administered as a powder-in-capsule once daily for 14 days immediately before breakfast, in healthy volunteers.
  Arms: 100 mg PF-05175157 or Placebo QD
Drug: PF-05175157 or Placebo — One oral dose of PF-05175157 or placebo is administered as a powder-in-capsule once daily for 14 days immediately before breakfast, in healthy volunteers.
  Arms: 200 mg PF-05175157 or Placebo QD
Drug: PF-05175157 or Placebo — One oral dose of PF-05175157 or placebo is administered as a powder-in-capsule twice daily for 14 days, immediately before breakfast and dinner, in healthy volunteers.
  Arms: 100 mg PF-05175157 or Placebo BID
Drug: PF-05175157 or Placebo — One oral dose of PF-05175157 or placebo is administered as a powder-in-capsule once (or twice) daily for 14 days, immediately before breakfast (and dinner), in patients with type 2 diabetes.
  Arms: xxx mg PF-05175157

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of PF-05175157 in healthy volunteers and patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.
* In addition, subjects must have normal pulmonary function tests and normal ocular examination.
* Body Mass Index (BMI) of 25.5 - 35.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Women must be of non-childbearing potential.
* Subjects with type 2 diabetes: HbA1c ≥7.0% and ≤10.0% if on metformin only, and ≥6.5% and ≤9.0% if patient requires to be washed-off an SU or DPP-4i.
* For subjects with type 2 diabetes, due to possible effects on disposition, CYP P450 3A4/5 and 2D6 substrates should not be co-administered with study medications.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic seasonal allergies at time of dosing).
* Evidence or history of any chronic ongoing or current pulmonary disease.
* History of smoking in the past 5 years and a history of smoking more than 10 pack years, or history or evidence of habitual use of other (non smoked) tobacco or nicotine containing products within 3 months of Screening, or positive cotinine test at Screening or Day -3.
* Active ocular disease including infection, glaucoma, seasonal allergies, dry eye symptoms or retinal/optic nerve disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Miami Research Associates, South Miami, Florida
  - MRA Clinical Research, South Miami, Florida
  - Pulmonary Physicians of South Florida, South Miami, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731007&StudyName=A%20Study%20of%20PF-05175157%20in%20Healthy%20Volunteers%20and%20Type%202%20Diabetic%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo - Healthy and Overweight Participants (HOV): HOV participants administered orally matched placebo capsules once daily (QD) for 14 days
- Placebo - Type 2 Diabetes Mellitus Participants (T2DM): T2DM participants administered orally matched placebo capsules QD for 14 days
- PF-05175157 30 mg QD - HOV: HOV participants administered orally 30 milligram (mg) capsules of PF-05175157 QD for 14 days
- PF-05175157 100 mg QD - HOV: HOV participants administered orally 100 mg capsules of PF-05175157 QD for 14 days
- PF-05175157 200 mg QD - HOV: HOV participants administered orally 200 mg capsules of PF-05175157 QD for 14 days
- PF-05175157 100 mg BID - HOV: HOV participants administered orally 100 mg capsules of PF-05175157 twice daily (BID) for 14 days
- PF-05175157 200 mg QD - T2DM: T2DM participants administered orally 200 mg capsules of PF-05175157 QD for 14 days
Period: Overall Study
Arm/Group | Placebo - Healthy and Overweight Participants (HOV) | Placebo - Type 2 Diabetes Mellitus Participants (T2DM) | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Started | 12 | 5 | 9 | 9 | 9 | 9 | 11
Completed | 12 | 5 | 9 | 9 | 8 | 9 | 10
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo - HOV: HOV participants administered orally matched placebo capsules QD for 14 days
- Placebo - T2DM: T2DM participants administered orally matched placebo capsules QD for 14 days
- PF-05175157 30 mg QD - HOV: HOV participants administered orally 30 mg capsules of PF-05175157 QD for 14 days
- PF-05175157 100 mg QD -HOV: HOV participants administered orally 100 mg capsules of PF-05175157 QD for 14 days
- PF-05175157 200 mg QD - HOV: HOV participants administered orally 200 mg capsules PF-05175157 QD for 14 days
- PF-05175157 100 mg BID - HOV: HOV participants administered orally 100 mg capsules of PF-05175157 BID for 14 days
- Total: Total of all reporting groups
Arm/Group | Placebo - HOV | Placebo - T2DM | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD -HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM | Total
Number analyzed (Participants) | 12 | 5 | 9 | 9 | 9 | 9 | 11 | 64
Age, Customized [Number; unit: participants]
  18 to 44 years | 9 | 2 | 9 | 7 | 8 | 7 | 2 | 44
  45 to 64 years | 3 | 3 | 0 | 2 | 1 | 2 | 9 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
  Male | 12 | 4 | 9 | 9 | 9 | 9 | 9 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to PF-05175157 was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: 2 weeks
Population: Safety Analysis Set: all participants who received at least 1 dose of study medication (PF-05175157 or placebo).
Measure: Number; unit: participants
Arm/Group | Placebo - HOV | Placebo - T2DM | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Number analyzed (Participants) | 12 | 5 | 9 | 9 | 9 | 9 | 11
participants
  AEs | 2 | 2 | 1 | 1 | 2 | 5 | 3
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Hour 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 1 and 14; at Hour 0 (pre-dose), 3.5, 12 hours post-dose for Day 4, 7 and 11
Population: Pharmacokinetic Concentration (PKC) Analysis Population: all enrolled participants who received at least 1 dose of PF-05175157 and had at least 1 concentration value reported. Number of Participants Analyzed (N): number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Arm/Group | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Number analyzed (Participants) | 9 | 8 | 8 | 9 | 10
micrograms per milliliter (µg/mL) | 3.07 (0.28) | 7.52 (2.87) | 21.75 (4.44) | 15.18 (2.11) | 23.26 (4.43)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 2
Population: Pharmacokinetic Parameter (PKP) Analysis Population: all enrolled participante who received at least 1 dose of PF05175157 and had at least 1 PKP of interest calculated;Number of Participants Analyzed (N): number of participants with evaluable data
Measure: Median (Full Range); unit: hours (hrs)
Arm/Group | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Number analyzed (Participants) | 9 | 8 | 8 | 9 | 10
hours (hrs) | 4.00 [1.00 to 4.00] | 1.00 [1.00 to 6.00] | 4.00 [3.00 to 4.00] | 3.00 [3.00 to 4.00] | 4.00 [2.00 to 6.00]

4. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Time Frame: as for outcome 2
Population: PKP analysis population; Participants Analyzed (N): number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: µg times (*)hr divided by mL (µg *hr/mL)
Arm/Group | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Number analyzed (Participants) | 9 | 8 | 8 | 9 | 10
µg times (*)hr divided by mL (µg *hr/mL) | 32.86 (4.01) | 90.50 (33.40) | 255.9 (36.98) | 125.6 (16.73) | 282.6 (66.21)

5. Secondary Outcome: Accumulation Ratio for Area Under the Concentration-Time Curve (Rˇac, AUC)
Description: Rˇac for the AUC is defined as AUC (τ, single dose [ss]) / AUC (τ, multiple dose [sd]).
Time Frame: as for outcome 2
Population: PKP analysis population; Participants Analyzed (N): number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Number analyzed (Participants) | 9 | 8 | 8 | 9 | 10
ratio | 1.39 (0.11) | 1.01 (0.34) | 1.47 (0.22) | 2.53 (0.76) | 1.54 (0.22)

6. Secondary Outcome: Renal Clearance (CLr)
Description: CLr is the amount of unchanged drug excreted in the participants urine from time zero to end of dosing interval.
Time Frame: as for outcome 2
Population: PKP analysis population; Participants Analyzed (N): number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Number analyzed (Participants) | 9 | 8 | 8 | 9 | 10
mL/min | 5.48 (1.25) | 5.30 (1.42) | 4.57 (1.83) | 5.93 (1.86) | 5.42 (1.38)

7. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: It was not possible to calculate data for half-life as the calculation required the slope of terminal elimination phase and the PK sampling was insufficient to characterize the terminal elimination phase, which is needed for the calculation of the half-life.
Arm/Group | Placebo - HOV | Placebo - T2DM | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Urinary Recovery
Description: Percentage of PF-05175157 excreted unchanged in urine over the dosing interval.
Time Frame: as for outcome 2
Population: PKP analysis population; Participants Analyzed (N): number of participants with evaluable data
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Number analyzed (Participants) | 9 | 8 | 8 | 9 | 10
percentage | 35.59 (7.78) | 27.30 (8.14) | 33.75 (9.53) | 43.60 (10.72) | 44.31 (7.79)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo - HOV | Placebo - T2DM | PF-05175157 30 mg QD - HOV | PF-05175157 100 mg QD - HOV | PF-05175157 200 mg QD - HOV | PF-05175157 100 mg BID - HOV | PF-05175157 200 mg QD - T2DM
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5 | 0/9 | 0/9 | 0/9 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 2/12 | 2/5 | 1/9 | 1/9 | 2/9 | 5/9 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - HOV (N=12) | Placebo - T2DM (N=5) | PF-05175157 30 mg QD - HOV (N=9) | PF-05175157 100 mg QD - HOV (N=9) | PF-05175157 200 mg QD - HOV (N=9) | PF-05175157 100 mg BID - HOV (N=9) | PF-05175157 200 mg QD - T2DM (N=11)
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival irritation (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.